CLINICAL TRIAL: NCT02061215
Title: Effects of Age on Immune Risk Profile in CMV Seropositive Kidney Transplant Recipients After Release From CMV Prophylaxis
Brief Title: Study of CMV in Kidney Transplant Recipients
Status: Terminated | Type: Observational
Why Stopped: PI halted study
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0742-13-EP
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: CMV Viral Loads in Seropositive Renal Transplant Recipients
Keywords: CYTOF; CMV; PCR; HLA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- recipients aged 20-40: CMV viral load
  Interventions: Other: CMV viral load
- recipients older than 60: CMV viral load
  Interventions: Other: CMV viral load

INTERVENTIONS:
Other: CMV viral load

SUMMARY:
Using novel CYTOF technology to measure a wide array of innate and adaptive cell proportions and cytokine levels, we plan a pilot study in old (>/=60 years) and young (20-40 years) renal transplant recipients who are cytomegalovirus (CMV) seropositive (regardless of donor serology). Viral load measurements will be performed at baseline prior to transplant (within 1 week),and then at 3, 7 and 10 months after transplant. It is expected that the patient will receive anti-CMV prophylaxis until 6 months post-transplant, so the latter two time points will reflect responses after "release" from antiviral suppression. Each patient will serve as their own control, with comparisons made between measurements at baseline and then at each timepoint. In addition, clinical data will be collected at the time points indicated, particularly renal function and the presence/absence of acute rejection.

DETAILED DESCRIPTION:
Using novel CYTOF technology to measure a wide array of innate and adaptive cell proportions and cytokine levels, we plan a pilot study in old (>/=60 years) and young (20-40 years) renal transplant recipients who are CMV seropositive (regardless of donor serology). Viral load measurements will be performed at baseline prior to transplant (within 1 week),and then at 3, 7 and 10 months after transplant. It is expected that the patient will receive anti-CMV prophylaxis until 6 months post-transplant, so the latter two time points will reflect responses after "release" from antiviral suppression. Each patient will serve as their own control, with comparisons made between measurements at baseline and then at each timepoint.

Blood from 10 patients in each age group will be studied, to collect virologic and immune response data:

* CYTOF (broad array of measurements)
* Tetramer assays (requires recipient HLA type of A1, A2, B7)
* CMV viral load PCR
* Response to pneumococcal antigens and inactivated influenza virus

In addition, clinical data will be collected at the time points indicated,particularly renal function and the presence/absence of acute rejection.

ELIGIBILITY:
Inclusion Criteria:

1. Adults young age 20-40 years and old >/= 60 years
2. Anticipate renal transplant within 2 weeks
3. CMV sero-positive renal transplant recipients
4. HLA type of A1, A2, B7 of recipient

Exclusion Criteria:

1. Pediatric recipients
2. Multi-organ transplant recipients
3. Highly sensitized (antigen level) recipients
4. Prior organ transplant recipients
5. Patients who do not wish to participate in study, or who cannot consent to research
6. Patients with active CMV infection
7. Seronegative
8. HLA Type of organ recipient not corresponding to A1,A2, B7

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recipients of renal transplants at the University of Nebraska Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07-14 (Actual); Study Completion 2015-07-14 (Actual)

PRIMARY OUTCOMES:
CMV viral loads in younger seropositive kidney transplant recipients before transplant, during treatment and after therapy | 1 year
  CMV viral loads in younger (age 20-40) seropositive kidney transplant recipients before renal transplant, during treatment with anti-viral therapy, and after release from therapy
CMV viral loads in older seropositive kidney transplant recipients before transplant, during treatment and after therapy | 1 year
  CMV viral loads in older (age >/= 60) seropositive kidney transplant recipients before renal transplant, during treatment with anti-viral therapy, and after release from therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Maskin, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States